CLINICAL TRIAL: NCT01383655
Title: The Efficacy of Intravenous Magnesium in Acute Wheezy Bronchitis in Small Children - a Randomized, Controlled Study
Brief Title: Intravenous Magnesium in Wheezy Bronchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Marjo Renko, docent, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVMg135/2010
Record Dates: First submitted 2011-06-06; First posted 2011-06-28 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Wheezy Bronchitis
Keywords: wheezy bronchitis; asthma; rhinovirus; magnesium
MeSH Terms: conditions — Bronchiolitis; Asthma | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium (Experimental): i.v. magnesium infusion 40mg/kg in 20 min
  Interventions: Drug: Magnesium Sulfate
- Placebo (Placebo Comparator): i.v. 0.9 % NaCl
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium Sulfate — i.v. magnesium 40mg/kg in 20 min
  Arms: Magnesium
Drug: Placebo — NaCl
  Arms: Placebo

SUMMARY:
In infants and toddlers wheezy bronchitis is a common viral disease. To relieve wheezing symptoms bronchodilators or corticosteroids are commonly used but the efficacy is not always satisfactory.

The purpose of this trial is to investigate the effectiveness of iv-magnesium in the treatment of moderate or severe bronchial obstruction associated with viral infection in small children.

The study population will include the children attending the Pediatric Emergency Department of Oulu University Hospital because of respiratory infection and bronchial obstruction that is not relieved with conventional treatment. After written consent from the parents, the children will be randomized to get either intravenous magnesium sulfate or isotonic NaCl. The primary outcome is RDAI (Respiratory Distress Assessment Instrument) scoring six hours from the infusion. Secondary endpoints are RDAI scoring and oxygen saturation at other time points and length of hospital stay.

The sample size is 64 children at the age of 6 months to 4 years.

If iv-magnesium is effective in relieving viral infection associated bronchial obstruction, that would be an important addition to the treatment of this common disease.

DETAILED DESCRIPTION:
In infants and toddlers wheezy bronchitis is a common viral disease. To relieve wheezing symptoms bronchodilators or corticosteroids are commonly used but the efficacy is not always satisfactory.

Intravenous infusion of magnesium sulfate has been proven to be efficacious and safe for the treatment of acute asthma attacks in adults and school-aged children. The purpose of this trial is to investigate the effectiveness of iv-magnesium in the treatment of moderate or severe bronchial obstruction associated with viral infection in small children.

The study population will include the children attending the Pediatric Emergency Department of Oulu University Hospital because of respiratory infection and bronchial obstruction that is not relieved with conventional treatment. After written consent from the parents, the children will be randomized to get either intravenous magnesium sulfate or isotonic NaCl. The primary outcome is RDAI (Respiratory Distress Assessment Instrument) scoring six hours from the infusion. Secondary endpoints are RDAI scoring and oxygen saturation at other time points and length of hospital stay.

The sample size is 64 children at the age of 6 months to 4 years.

If iv-magnesium is effective in relieving viral infection associated bronchial obstruction, that would be an important addition to the treatment of this common disease.

ELIGIBILITY:
Inclusion Criteria:

* age 0.5 - 4 years
* wheezy bronchitis
* RDAI > 6 after conventional treatment

Exclusion Criteria:

* prematurity
* congenital heart disease
* immune deficiency

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2011-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
RDAI score | 6h

SECONDARY OUTCOMES:
saturation | 6h
RDAI | 2h
saturation | 2h
length of hospital stay | length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Marjo Renko, MD, Study Chair — University of Oulu, Department of Pediatrics
Locations (1):
- Department of Pediatrics, Oulu University Hospital, Oulu, Oulu, Finland

REFERENCES:
- [Derived] Pruikkonen H, Tapiainen T, Kallio M, Dunder T, Pokka T, Uhari M, Renko M. Intravenous magnesium sulfate for acute wheezing in young children: a randomised double-blind trial. Eur Respir J. 2018 Feb 7;51(2):1701579. doi: 10.1183/13993003.01579-2017. Print 2018 Feb. PMID 29437941